CLINICAL TRIAL: NCT05122039
Title: ProspectIve Cohort psoriASiS fOllow-up (PICASSO)
Acronym: PICASSO
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s64740
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Patient visits are planned at baseline and after 2.5, 5, 7.5 and 10 years. At all time-points clinical examination and parameters, anamnesis, clinical pictures and questionnaires will be completed. The following samples will be taken at all time-points:
  * Blood (serum, plasma, DNA)
  * Skin tape stripping (psoriatic and healthy skin)(mRNA-analysis)
  * Skin swabs (psoriatic and healthy skin)(skin microbiome)
  * Nails (DNA-analysis)
  * Faecal samples (faecal microbiome)
  * Saliva samples (mRNA-analysis, oral microbiome)
  * Urine samples (metabolomics)
  The following examinations are optional:
  * Skin biopsy
  * Hair sample
  * Carotid Intima Media thickness (ultra-sound)
  * Examination of the oral cavity
  * Ocular swab (ocular microbiome)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of the PICASSO-project is to facilitate future psoriasis-research in dermatology. This register biobank will enable us to perform research in the field of metabolomics, mRNA-expression, cardiovascular impact and the microbiome. The final aims are patient stratification, better insight in disease-evolution and improved understanding of markers that predispose to severe disease.

DETAILED DESCRIPTION:
The PICASSO-project is a prospective register with extensive biobanking in which patients with a recent onset of psoriasis (<3 years) can be enrolled. Participants are followed for a period of 10 years, with scheduled visits every 2.5 years. The same protocol is followed for every visit. The registry captures patient demographics, medical history (personal and family), details of psoriasis treatment (previous and current), physical examination, disease activity scores and PROMs. Some patients (substudy) will undergo ultra-sound to determine carotid intima media thickness. Biobanking in this project encompasses extensive biosampling of multiple tissues. It is not within the scope of this project to administer study medication: patients receive standard of care treatment as prescribed by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of Psoriasis since >3 years
* adults (70 years old or less) and children (>12 years old)
* willing and able to understand and sign the informed consent (plus legal representative in case of a minor)

Exclusion Criteria:

* unwilling or unable to understand and sign the informed consent
* disease duration longer than 3 years

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Psoriasis patients with disease duration less than three years, aged 12-70 years old at time of inclusion
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2032-10-19 (Estimated); Study Completion 2032-10-19 (Estimated)

PRIMARY OUTCOMES:
We hypothesize that metabolic state in early disease (<3 years of disease onset) is linked to and predictive of more severe course of psoriasis after five years. | 10 years
  To describe the presence/absence of metabolic syndrome (defined by clinical parameters and cut-off levels of associated adipokines (see section 'Background': ref 8-11)) in early disease, and link it to disease severity (eg. mild psoriasis (PASI 0.1-4); moderate psoriasis (PASI 4.1-9.9); severe psoriasis (PASI 10 and above OR receiving systemic treatment/biologics); BSA: mild to moderate (0.1-5%); moderate to severe (5 and above)). It is within the primary endpoint of this project to re-evaluate both MetS- and psoriasis-parameters after 2.5, 5, 7.5 and 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hillary, MD, Principal Investigator — Department of Dermatology, University Hospitals Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. Data on cohort-level will be published.